CLINICAL TRIAL: NCT05015426
Title: Phase 1/1b Trial of Donor γδ T--Cell Infusion for Treatment of Patients With Acute Myeloid Leukemia at High Risk of Relapse After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Gamma Delta T-cell Infusion for AML at High Risk of Relapse After Allo HCT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20305; 9BC08 (Other Grant/Funding Number: Florida Department of Health)
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level -1 (Experimental): Dose Level -1 may be used as a de-escalation dose level due to Dose Limiting Toxicities (DLTs) from Dose Level 1
  Participants will receive 1.0 x 106 cells/kg (0.75-1.25 x 106 cells/kg) Artificial Antigen Presenting Cell (AAPC)-expanded donor T-cells administered as a single infusion
  Interventions: Biological: Gamma Delta T-Cell Infusion
- Dose Level 1 (Experimental): Participants will receive 5.0 x 106 cells/kg (3.75-6.25 x 106 cells/kg) Artificial Antigen Presenting Cell (AAPC)-expanded donor T-cells administered as a single infusion
  Interventions: Biological: Gamma Delta T-Cell Infusion
- Dose Level 2 (Experimental): Participants will receive 2.5 x 107 cells/kg (1.875-3.125 x 107 cells/kg) Artificial Antigen Presenting Cell (AAPC)-expanded donor T-cells administered as a single infusion
  Interventions: Biological: Gamma Delta T-Cell Infusion
- Dose Level 3 (Experimental): Participants will receive 1.0 x 108 cells/kg (0.75-1.25 x 108 cells/kg) Artificial Antigen Presenting Cell (AAPC)-expanded donor T-cells administered as a single infusion
  Interventions: Biological: Gamma Delta T-Cell Infusion
- Treatment at Maximum Tolerated Dose (Experimental): Participants will receive Artificial Antigen Presenting Cell (AAPC)-expanded donor T-cells at the dose determined to be the Maximum Tolerated Dose, administered as a single infusion
  Interventions: Biological: Gamma Delta T-Cell Infusion

INTERVENTIONS:
Biological: Gamma Delta T-Cell Infusion — Donor cells will be processed in a laboratory, where T-cell subtype called γδ (gamma delta) T-cells will be isolated and expanded in number. These T-cells expanded in a laboratory will be infused in participants who are otherwise at high risk of AML recurrence after alloHCT.

SUMMARY:
The purposes of the study are to determine the maximum tolerated dose (MTD) and effectiveness of Artificial Antigen Presenting Cell (AAPC)-expanded donor T-cells administered as a single infusion after an allogeneic hematopoietic cell transplant (alloHCT) to treat patients with Acute Myeloid Leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 and 75 years of age undergoing allogeneic hematopoietic stem cell transplantation (alloHCT) or the treatment ELN 2017 adverse risk AML
* Have < 5% blasts in bone marrow by morphology at the time of transplantation. Patients with pre-alloHCT or post-alloHCT flow cytometric or molecular evidence of MRD are allowed
* Karnofsky performance status (KPS) ≥ 70% during the study screening.
* Free of symptomatic congestive heart failure or uncontrolled arrhythmia
* Adequate organ function as defined per protocol
* Negative serum pregnancy test
* Note: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for at least 30 days following study treatment (T-cell infusion); should a woman subject or female partner of a male subject become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Current use of concomitant systemic glucocorticoid at the time of γδ T-cell infusion for any reason will not be allowed in order to avoid their immunosuppressive effects on γδ T-cell function.
* Active grade II-IV acute GVHD (patients with prior GVHD should be off prednisone for at least 14 days prior to infusion of the study cell product).
* Uncontrolled serious infection.
* Morphologic relapse of leukemia at any timepoint after HCT.
* Active central nervous system malignancy.
* Pregnancy or lactation.
* Treatment with another investigational drug or other intervention within 14 days of T-cell infusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 12 months
  Maximum Tolerated Dose will be determined by testing increasing doses of AAPC-expanded donor γδ T-cells.
Dose Expansion: Leukemia Free Survival | Up to 12 months
  Leukemia-free survival is defined as the time from the date of start of treatment to the date of relapse of AML or death from any cause

SECONDARY OUTCOMES:
Number of Participants with Graft Versus Host Disease (GVHD) | at 6 weeks
  Number of participants with grade II-IV and III-IV acute GVHD within 6 weeks after infusion of Gamma T cells
Overall Survival (OS) | Up to 12 months
  The length of time from start of treatment to death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Nelli Bejanyan, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States